CLINICAL TRIAL: NCT06331624
Title: Biomarker Modulation and the Inhibition of Natural Killer Type 1 (NKT1) Cells by Oral GRI-0621 in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Biomarker Modulation and the Inhibition of NKT1 Cells by Oral GRI-0621 in Patients With IPF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GRI Bio Operations, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GRI-0621-IPF-02
Record Dates: First submitted 2024-02-01; First posted 2024-03-26 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Idiopathic Pulmonary Fibrosis; IPF
Keywords: Idiopathic Pulmonary Fibrosis; IPF; Biomarker Modulation; Inhibition of Natural Killer Type 1 (NKT1) Cells; NKT Cells; GRI-0621; Tazarotene
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — tazarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GRI-0621 (Experimental): GRI-0621 (tazarotene) 4.5mg, administered orally once daily (QD)
  Interventions: Drug: Tazarotene (GRI-0621)
- Placebo (Experimental): Placebo 4.5mg, administered orally once daily (QD)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tazarotene (GRI-0621) — Oral 4.5mg soft gel capsule
  Arms: GRI-0621
Drug: Placebo — Oral 4.5mg soft gel capsule
  Arms: Placebo

SUMMARY:
This is a Phase 2a, randomized, double-blind, multi-center, placebo-controlled, parallel-design, 2-arm study. Approximately 36 subjects with IPF will be randomized in a 2:1 ratio for GRI-0621 4.5mg or Placebo. GRI-0621 dose of 4.5mg will be compared with placebo following once daily oral administration for 12 weeks.

Concurrently, a Sub-Study will be conducted, examining the number and activity of NKT cells in BAL, for up to 12 eligible subjects (across various centers).

An early-stage patient variability assessment will be completed when 12 subjects have completed 2 weeks of treatment. Followed by an interim analysis performed when 24 subjects complete 6 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 40 through 85 years of age, inclusive.
2. Confirmed diagnosis of IPF with clinical features consistent with the current clinical practice guidelines for IPF.
3. FVC > 50% predicted value within 4 weeks of Screening.
4. FEV1/FVC ratio > 0.65 within 4 weeks of Screening.
5. Diffusion capacity for carbon monoxide corrected for hemoglobin (DLCOc) > 30%predicted value within 4 weeks of Screening.
6. Life expectancy of at least 12 months.
7. Willing and able to follow the study required visits and assessments. For Sub-Study subjects, willing and able to undergo BAL procedures at Screening and at Week 12.
8. Willing and able to provide written informed consent prior to study-related procedures.

Exclusion Criteria:

1. Initiation of any approved or investigational IPF therapy or oral corticosteroids (> 10 mg/day) within 4 weeks of Screening. Subjects already on approved IPF therapies must remain on their current medication from Screening until the last study visit.
2. High resolution computerized tomography (HRCT) pattern showing emphysema more than the extent of fibrosis of the lung area within 12 months of Screening.
3. Acute exacerbation of IPF within 6 months of Screening (Collard et al., 2016).
4. Requiring supplemental O2 > 4 liters/min to maintain peripheral arterial O2 saturation (SpO2) > 88% at rest. O2 saturation at screening or baseline that is < 88% at rest.
5. Any condition with unacceptable risk for bronchoscopy (for Sub-Study subjects only).
6. Current or recent history of clinically significant medical condition, laboratory abnormality, or illness that could place the subject at risk or compromise the quality of the study data as determined by the Investigator.
7. Significant coronary artery disease (i.e., myocardial infarction within 6 months or unstable angina within 1 month of Screening).
8. An upper or lower respiratory tract infection, presence of or suspected emphysema, within 4 weeks of Screening.
9. Eye exam indicating night blindness within 6 months of Screening, or at Screening.
10. Bone Mineral Density t-score of -4.0 (severe osteoporosis) within 6 months of Screening, or at Screening.
11. Screening QT of >450 for men and >470 for women.
12. History of renal impairment as deemed clinically relevant by the investigator OR eGFR <60ml/min/1.73m2 within 60 days of Screening and a Screening eGFR of <60ml/min/1.73m2.
13. History of hepatic impairment as deemed clinically relevant by the investigator OR ALT or AST >2 x ULN OR moderate and severe hepatic impairment as defined using the Child-Pugh scoring system (i.e., Child-Pugh B and C).
14. A history of hypertriglyceridemia (documented TG of >2.0mmol/L at Screening); a history of pancreatitis from any cause; uncontrolled dyslipidemia with LDL-c >4.9mmol/L and an HDL-c <1.3 mmol/L for women and <1.0 for men, despite optimized treatment.
15. Use of moderate or strong inhibitors of CYP2C8 (e.g. gemfibrazol, trimethoprim, clopidogrel) or inducers of CYP2C8 (e.g. rifampin) from 7 days or 5 half-lives, whichever is longer, before the first administration of GRI-0621 until cessation of GRI-0621 administration.
16. Subjects who report any active suicidal ideation (SI) or behavior (SB) (i.e. Columbia Suicide Severity Rating Scale (C-SSRS) scores 4 or greater for SI and any positive scores for SB) during Screening or any past history thereof.
17. Current smoker (i.e., use of tobacco products within the last 3 months) of Screening.
18. Current or recent history of drug or alcohol abuse within 12 months of Screening.
19. Participation in any other investigational drug study within 4 weeks of Screening or within 5 times the elimination half-life of an investigational drug.
20. Females who are pregnant or breastfeeding, or if of child-bearing potential unwilling to practice two highly effective forms of contraception for at least 1 month prior to initiation of the study drug, during the study, and for 1 month after discontinuing the study drug (e.g., abstinence, intrauterine device or system, combination of barrier and spermicide, hormonal contraceptive, surgical sterilization, or male partner sterilization).
21. Males, if sexually active, unwilling to practice two highly effective forms of contraception during the study (e.g., condom, or surgical sterilization).
22. History of hypersensitivity or intolerance to oral tazarotene.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of oral GRI-0621 | 12 Weeks
  General overall safety and tolerability of oral GRI-0621 as compared to placebo will be assessed by evaluating the following safety parameters:
  * Adverse events (occurrence and type)
  * Clinical Laboratory Measurements (normal/abnormal)
  * Vital signs (normal/abnormal)

SECONDARY OUTCOMES:
Change from baseline biomarkers | 12 Weeks
  Change from baseline in biomarkers (PRO-C3, PRO-C6, C1M, C3M, C6M, VICM, CPa9-HNE, PRO-C4, PRO-C5, CTX-III, ELP-3, C4Ma3)
Plasma concentrations of GRI-0621 | 12 Weeks
  Pharmacokinetic analysis
Pharmacodynamics of GRI-0621 in blood (Study Population) | 6 Weeks and 12 Weeks
  Measure of NKT1 cell activation inhibition in blood
Pharmacodynamics of GRI-0621 in BAL fluid (Optional Sub-Study) | 12 Weeks
  Measure of NKT1 cell activation inhibition from bronchoalveolar lavage (BAL) fluid

OTHER OUTCOMES:
Exploratory - Pulmonary Function | 6 Weeks and 12 Weeks
  Effect of GRI-0621 on pulmonary function (FEV1, FVC, and FEV1/FVC ratio) at baseline and after 6 weeks and 12 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (5):
  - Newport Native MD, Inc., Newport Beach, California
  - Mayo Clinic, Jacksonville, Florida
  - Montefiore Medical Center, The Bronx, New York
  - Southeastern Research Center, Winston-Salem, North Carolina
  - MUSC Pulmonary Research, Charleston, South Carolina
- Australia (3):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Concord General Repatriation Hospital, Concord, New South Wales
  - St. George Hospital, Kogarah, New South Wales
- United Kingdom (8):
  - Royal Infirmary Edinburgh, Edinburgh, Scotland
  - University Hospital Birmingham, Queen Elizabeth Hospital, Birmingham
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - Royal Devon and University Healthcare NHS Foundation Trust, Exeter
  - University College London Hospitals, London
  - Western Health and Social Care Trust (WHSCT), Londonderry
  - Norfolk & Norwich University Hospital, Norwich
  - Oxford University Hospitals NHS Foundation Trust, Oxford